CLINICAL TRIAL: NCT02485119
Title: An Open Label, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BAY94-9343 Given by Intravenous Infusion Every 3 Weeks (Q3W) in Japanese Subjects With Advanced Malignancies
Brief Title: Phase I Dose Escalation Study of BAY94-9343 Given by Intravenous Infusion Every 3 Weeks in Japanese Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15404
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Neoplasms
Keywords: BAY 94-9343; Anetumab ravtansine; ADC (Antibody Drug Conjugate); Phase I; Japan; solid cancers; Advanced, refractory solid tumors; mesothelin; endometrial; adenocarcinoma of lung; gastrointestinal, ovarian, pancreatic, cholangio, mesothelioma and triple negative breast cancers
MeSH Terms: conditions — Neoplasms; Adenocarcinoma of Lung; Mesothelioma; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY94-9343 (Experimental): Cohort 1: Safety, tolerability and PK of 4.5 mg/kg dose given Q3W. Proceeding to Cohort 2 or not will be decided based on both safety variables during Cycle 1 (21 days) of 3 to 6 subjects in Cohort 1 and PK obtained from Cycle 1 (at least Day 1 to Day 5).
  Cohort 2: Safety, tolerability and PK of 6.5 mg/kg dose given Q3W. Whether recruitment will be continued up to 9 subjects for Cohort 2 or not will be decided based on safety variables during Cycle 1 (21 days) of the first 3 subjects in Cohort 2. The safety and tolerability of 6.5 mg/kg will be assessed based on the data of 9 subjects during Cycle 1 in Cohort 2, and considering long term toxicity, the safety and tolerability of BAY94-9343 will be assessed all safety data by the end of 3 cycles in Cohort 2.
  Interventions: Drug: BAY94-9343

INTERVENTIONS:
Drug: BAY94-9343 — Cohort 1: 4.5 mg/kg of BAY 94-9343 at Q3W dose regimen. Cohort 2: 6.5 mg/kg of BAY 94-9343 at Q3W dose regimen.

SUMMARY:
The primary objectives of the Phase I study 15404 are to evaluate the safety, tolerability and pharmacokinetics of BAY94-9343 given once every 3 weeks in Japanese subjects with advanced, refractory solid tumors.

The secondary objectives are to investigate the efficacy, biomarkers and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects ≥ 20 years of age
* ECOG Performance Status of 0 to 1
* Life expectancy of at least 12 weeks
* Subjects with advanced, histologically or cytologically confirmed solid tumors, not amenable to any standard therapy, have no standard therapy available
* Subjects whose fresh or archival tumor tissues are available
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension according to RECIST criteria (Version 1.1 or modified version)
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Anticancer chemotherapy, experimental cancer therapy, or immunotherapy within 2 weeks of start of the first dose
* Impaired cardiac function or clinically significant cardiac disease (i.e., congestive heart failure (CHF) NYHA Class III or IV)
* Myocardial infarction or onset of unstable angina < 3 months prior to general screening
* Cardiac arrhythmias in the electrocardiogram that would interfere with QT/QTc interval measurement (LBBB (left bundle branch block), AV block, atrial fibrillation)
* QTc >470 ms, derived as the average of the 3 values measured by the ECG recorder's algorithm on the ECG triplicate
* LVEF (left ventricular ejection fraction) <50 %
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection
* Subjects with an active hepatitis B or C infection requiring treatment
* Personal or family history of Long QT Syndrome (LQTS)
* Subject with clinically significant eye disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-emergent Adverse Events (TEAEs) as a measure of safety and tolerability | Up to 9 weeks
Intensity of TEAEs acc. to NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v.4.03 | Up to 9 weeks
Cmax (maximum drug concentration in plasma after single dose administration ) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)
Cmax,norm (Cmax divided by dose (mg) per kg body weight) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)
Cmax/D (Cmax divided by dose (mg)) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)
AUC(0-tlast) (area under the plasma concentration vs time curve from time 0 to the last data point) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)
AUC(0-tlast)norm (AUC(0-tlast) divided by dose (mg) per kg body weight) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)
AUC(0-tlast)/D (AUC(0-tlast) divided by dose (mg)) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)
tmax (time to reach maximum drug concentration in plasma) for BAY94-9343, total antibody compound, DM4, metabolite DM4-Me | Cycle 1, 3 ,6: pre, 30, 60min, 1.5, 2, 3, 5, 8, 48, 96, 168 and 504 hours after the start of dosing; Cycle1,2 only: 336 hours; Cycle1 only: 24 hours (each cycle is 21 days)

SECONDARY OUTCOMES:
Tumor response based on RECIST (Response Evaluation Criteria in Solid Tumors) | Up to 9 weeks
Level of mesothelin expression using IHC (Immunohistochemistry) staining for the tumor tissue obtained from fresh or archival tumor tissue | Up to 9 weeks
Plasma levels of soluble mesothelin | Up to 9 weeks
Immunogenicity evaluation based on anti-BAY94-9343 antibody count | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Tyuo